CLINICAL TRIAL: NCT02761980
Title: A Phase 3, Double-blind, Randomized, Placebo-controlled, Full Factorial, Safety And Efficacy Study Comparing The Antipyretic Effects Of A Single Oral Dose Of Ibuprofen (Ibu) 250 Mg/ Acetaminophen (Apap) 500 Mg Caplets To Ibu 250 Mg And Apap 500 Mg Caplets In Healthy Male Volunteers With Fever Induced By An Endotoxin
Brief Title: A Study of Ibuprofen 250 mg / Acetaminophen 500 mg Comparing The Antipyretic Effects in Healthy Male Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B5061002; GEMINI IF (Other: Alias Study Number)
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Fever
Keywords: ibuprofen; acetaminophen; induced fever; fever
MeSH Terms: conditions — Fever | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ibuprofen 250 mg / Acetaminophen 500 mg (Experimental): Single dose of 2 caplets of Ibuprofen 125 mg / Acetaminophen 250 mg by mouth
  Interventions: Drug: Ibuprofen 250 mg / Acetaminophen 500 mg
- Ibuprofen 250 mg (Active Comparator): Single dose of 2 caplets of IBU 125 mg by mouth
  Interventions: Drug: Ibuprofen 250 mg
- Acetaminophen 500 mg (Active Comparator): Single dose of 1 APAP 500 mg caplet + 1 placebo caplet by mouth
  Interventions: Drug: Acetaminophen 500 mg
- Placebo (Placebo Comparator): Single dose of 2 caplets of Placebo by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen 250 mg / Acetaminophen 500 mg — Ibuprofen 250 mg / Acetaminophen 500 mg
  Other Names: IBU 250 / APAP 500
  Arms: Ibuprofen 250 mg / Acetaminophen 500 mg
Drug: Ibuprofen 250 mg — Ibuprofen 250 mg
  Other Names: IBU 250
  Arms: Ibuprofen 250 mg
Drug: Acetaminophen 500 mg — 1 APAP 500 mg caplet
  Other Names: APAP 500
  Arms: Acetaminophen 500 mg
Drug: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
This is a single dose study that will evaluate the efficacy and safety of a Fixed Dose Combination Ibuprofen 250 mg/ Acetaminophen 500 mg tablet in healthy male patients with fever. Results for the Fixed Dose Combination product will be compared to the individual components Ibuprofen 250 mg and Acetaminophen 500 mg and also compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects who, at the time of screening, are between 18 and 55 years of age, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests.
2. The subject must have a normal, stable body temperature at Screening and on Day 0. If the subject's oral temperature is not between 97.4°F and 98.8°F, then 2 additional oral temperature readings will be obtained within a 30 minute period. These 3 consecutive temperature readings must be between 97.4°F and 98.8°F, with the highest value within 0.4°F of the lowest temperature value.
3. Body Mass Index (BMI) of 17.5 to 37.0 kg/m2; and a total body weight 50 kg (110 lbs) at Screening.
4. The subject has demonstrably adequate veins, by visual inspection, for IV catheter insertion.

Exclusion Criteria:

1. Evidence or history of clinically significant laboratory abnormality, hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (excluding untreated, asymptomatic, seasonal allergies at the time of dosing) within the last 5 years that may increase the risk associated with study participation.
2. Subjects with any gastrointestinal disorders (eg, gastrectomy, tracheostomy, esophageal surgeries, short gut syndrome, peptic ulcer disease, known or suspected obstructive disease, previous gastrointestinal surgery, felinization of the esophagus, hypomotility of the gastrointestinal track) that could affect the absorption, metabolism, or excretion of the study medication or affect the results of the ingestible thermometer.
3. Subjects at risk for excessive bleeding.
4. Subjects with a history of nasal polyps, angioedema, or significant or actively treated bronchospastic disease.
5. Screening supine blood pressure ≤90 or ≥140 mm Hg (systolic) or ≤50 or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If blood pressure (BP) is ≤90 or ≥140 mm Hg (systolic) or ≤50 or ≥90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three consecutive BP values should be used to determine the subject's eligibility.
6. Screening supine 12 lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec at Screening and on Day 1 prior to RSE administration. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three consecutive QTc or QRS values should be used to determine the subject's eligibility.
7. The subject has a history of recurrent or acute or chronic infections of any type or any findings suggestive of occult infection, such as tuberculosis, sinusitis, urinary tract infection, respiratory tract or dental (abscess) infection, etc., or those with a positive QuantiFERON Tuberculosis, Hepatitis B surface antigen, Hepatitis C antibody, and/or Human immunodeficiency virus (HIV) test at Screening. Also excluded are subjects with frequent (more than 3 outbreaks per year), recurrent oral or genital herpes, recurrent herpes zoster, or any infection otherwise judged by the investigator to have the potential for exacerbation by participation in the study.
8. Subjects who have experienced cold/flu symptoms (ie, runny nose, cough, and/or fever) within 2 weeks prior to the first administration of study treatments.
9. Subjects with a reduction in heart rate to ≤50 beats per minute or deemed to be at high risk of syncope and/or hypotension per the clinical judgment of the investigator following a carotid sinus massage procedure.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 290 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Orleans Center for Clinical Research, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Smith W, Leyva R, Kellstein D, Arthur E, Cruz-Rivera M. Efficacy of a Fixed-Dose Combination of Ibuprofen and Acetaminophen Compared With Individual Monocomponents in Adult Male Subjects With Endotoxin-Induced Fever: A Randomized Controlled Trial. Clin Ther. 2021 Jul;43(7):1213-1227. doi: 10.1016/j.clinthera.2021.05.004. Epub 2021 Jul 23. PMID 34304913
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5061002&StudyName=A%20Phase%203%2C%20Double-blind%2C%20Randomized%2C%20Placebo-controlled%2C%20Full%20Factorial%2C%20Safety%20And%20Efficacy%20Study%20Comparing%20The%20Antipyretic%20Effects%20Of%20A%20Single%20Oral%20Dose%20Of%20Ibuprofen%20%28ibu%29%20250%20Mg%2F%20Acetaminophen%20%28apap%29%20500%20Mg%20Caplets%20To%20Ibu%20250%20Mg%20And%20Apap%20500%20Mg%20Caplets%20In%20Healthy%20Male%20Volunteers%20With%20Fever%20Induced%20By%20An%20Endotoxin
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5061002&StudyName=A+Phase+3%2C+Double-blind%2C+Randomized%2C+Placebo-controlled%2C+Full+Factorial%2C+Safety+And+Efficacy+Study+Comparing+The+Antipyretic+Effects+Of+A+Single+Oral+Dose+Of+Ibuprofen+%28ibu%29+250+Mg%2F+Acetaminophen+%28apap%29+500+Mg+Caplets+To+Ibu+250+Mg+And+Apap+500+Mg+Caplets+In+Healthy+Male+Volunteers+With+Fever+Induced+By+An+Endotoxin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, participants were administered at least 1 test dose of reference standard endotoxin (RSE) intravenously, based on their body weight before randomization, to induce pyrexia in them.
Groups:
- Placebo: Participants received placebo as single oral dose tablets during the treatment duration of 8 hours. Participants were discharged after completion of study treatment.
- Ibuprofen 250 mg+Acetaminophen 500 mg: Participants received single oral dose of a fixed dose combination of ibuprofen 250 milligram (mg) and acetaminophen 500 mg tablets during the treatment duration of 8 hours. Participants were discharged after completion of study treatment.
- Ibuprofen 250 mg: Participants received single oral dose of ibuprofen 250 mg tablet during the treatment duration of 8 hours. Participants were discharged after completion of study treatment.
- Acetaminophen 500 mg: Participants received single oral dose of acetaminophen 500 mg tablet during the treatment duration of 8 hours. Participants were discharged after completion of study treatment.
Period: Overall Study
Arm/Group | Placebo | Ibuprofen 250 mg+Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 500 mg
Started | 29 | 87 | 87 | 87
Completed | 25 | 80 | 81 | 81
Not Completed | 4 | 7 | 6 | 6
Not completed — Adverse Event | 4 | 6 | 5 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received study medication.
Groups:
- Ibuprofen 250 mg+Acetaminophen 500 mg: Participants received single oral dose of a fixed dose combination of ibuprofen 250 mg and acetaminophen 500 mg tablets during the treatment duration of 8 hours. Participants were discharged after completion of study treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen 250 mg+Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 500 mg | Total
Number analyzed (Participants) | 29 | 87 | 87 | 87 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (7.97) | 33.4 (10.54) | 32.3 (10.19) | 32.6 (9.99) | 32.4 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 29 | 87 | 87 | 87 | 290
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 4 | 3 | 13
  Not Hispanic or Latino | 27 | 83 | 83 | 84 | 277
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 10 | 20 | 12 | 47
  White | 21 | 72 | 65 | 69 | 227
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 2 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Sum of Temperature Difference (WSTD) From 0 to 8 Hours
Description: WSTD 0-8 was defined as time-weighted sum of temperature differences over 8 hours, weighted by time elapsed between each 2 consecutive time points post treatment (10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110 minutes, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5 and 8 hours). Temperature difference was defined as baseline temperature (at 0 hour) minus the post-baseline temperature at each time point up to 8 hours (10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110 minutes, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5 and 8 hours).
Time Frame: 0 to 8 hours post-dose
Population: Modified intent to treat (mITT) population included all randomized participants who were dosed with the study medication and RSE per procedures specified in protocol post amendment 4 and had a baseline assessment. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: degrees fahrenheit
Arm/Group | Placebo | Ibuprofen 250 mg+Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 500 mg
Number analyzed (Participants) | 27 | 81 | 83 | 82
degrees fahrenheit | 9.28 (6.395) | 12.54 (5.519) | 11.09 (6.355) | 12.39 (6.278)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg+Acetaminophen 500 mg; Treatment difference and 95 percent (%) confidence interval (CI) were based on Least Square Mean (LSM) from analysis of covariance (ANCOVA) with treatment, and covariates time from the first RSE full dose to randomization, and baseline temperature; Test type: Superiority; p = 0.002, ANCOVA; LSM difference = 3.14, 95% CI 2-sided [1.13 to 5.15]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Ibuprofen 250 mg; Treatment difference and 95 % CI were based on LSM from ANCOVA with treatment, and covariates time from the first RSE full dose to randomization, and baseline temperature; Test type: Superiority; p = 0.210, ANCOVA; LSM difference = 0.91, 95% CI 2-sided [-0.52 to 2.33]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Acetaminophen 500 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.280, ANCOVA; LSM difference = 0.79, 95% CI 2-sided [-0.64 to 2.21]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; Test type: Superiority — Treatment difference and 95 % CI were based on LSM from ANCOVA with treatment, and covariates time from the first RSE full dose to randomization, and baseline temperature; p = 0.030, ANCOVA; LSM difference = 2.23, 95% CI 2-sided [0.22 to 4.25]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 500 mg; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.023, ANCOVA; LSM difference = 2.35, 95% CI 2-sided [0.33 to 4.37]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 500 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.864, ANCOVA; LSM difference = -0.12, 95% CI 2-sided [-1.54 to 1.29]

2. Secondary Outcome: Time Weighted Sum of Temperature Differences (WSTD) From Baseline Through Hours 2, 4 and 6
Description: WSTD 0-2, 0-4 and 0-6 was defined as time-weighted sum of temperature differences over each specified time interval (0-2 hour, 0-4 hour and 0-6 hour), weighted by time elapsed between each 2 consecutive time points post treatment (10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110 minutes, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6 hour), within each time interval. Temperature difference was defined as baseline temperature (at 0 hour) minus the post-baseline temperature at each time point within each specified time interval: 1) 0-2 hour (20, 30, 40, 50, 60, 70, 80, 90, 100, 110 minutes) , 2) 0-4 hour (10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110 minutes, 2, 2.5, 3, 3.5, 4 hour), 3) 0-6 hour (10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110 minutes, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6 hour).
Time Frame: 0 to 2 hours postdose, 0 to 4 hours postdose, 0 to 6 hours postdose
Population: mITT population included all randomized participants who were dosed with the study medication and RSE per procedures specified in protocol post amendment 4 and had a baseline assessment. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: degrees fahrenheit
Arm/Group | Placebo | Ibuprofen 250 mg+Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 500 mg
Number analyzed (Participants) | 27 | 81 | 83 | 82
degrees fahrenheit
  WSTD 0-2 | -0.42 (1.827) | 0.48 (1.829) | -0.19 (1.856) | 0.21 (1.732)
  WSTD 0-4 | 1.79 (3.443) | 3.69 (3.152) | 2.61 (3.345) | 3.41 (3.173)
  WSTD 0-6 | 5.26 (4.833) | 7.95 (4.245) | 6.65 (4.788) | 7.65 (4.604)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg+Acetaminophen 500 mg; WSTD 0-2 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.004, ANCOVA; LSM difference = 0.90, 95% CI 2-sided [0.29 to 1.51]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Ibuprofen 250 mg; WSTD 0-2 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.078, ANCOVA; LSM difference = 0.39, 95% CI 2-sided [-0.04 to 0.82]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Acetaminophen 500 mg; WSTD 0-2 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.172, ANCOVA; LSM difference = 0.30, 95% CI 2-sided [-0.13 to 0.74]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; WSTD 0-2 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.098, ANCOVA; LSM difference = 0.51, 95% CI 2-sided [-0.10 to 1.13]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 500 mg; WSTD 0-2 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.054, ANCOVA; LSM difference = 0.60, 95% CI 2-sided [-0.01 to 1.21]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 500 mg; WSTD 0-2 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.692, ANCOVA; LSM difference = -0.09, 95% CI 2-sided [-0.52 to 0.34]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg+Acetaminophen 500 mg; WSTD 0-4 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p < 0.001, ANCOVA; LSM difference = 1.87, 95% CI 2-sided [0.86 to 2.88]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Ibuprofen 250 mg; WSTD 0-4 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.094, ANCOVA; LSM difference = 0.61, 95% CI 2-sided [-0.10 to 1.33]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Acetaminophen 500 mg; WSTD 0-4 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.217, ANCOVA; LSM difference = 0.45, 95% CI 2-sided [-0.27 to 1.17]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; WSTD 0-4 hours; Test type: Superiority; p = 0.015, ANCOVA — Treatment difference and 95 % CI were based on LSM from ANCOVA with treatment, and covariates time from the first RSE full dose to randomization, and baseline temperature; LSM difference = 1.26, 95% CI 2-sided [0.24 to 2.27]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 500 mg; WSTD 0-4 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.006, ANCOVA; LSM difference = 1.42, 95% CI 2-sided [0.40 to 2.44]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 500 mg; WSTD 0-4 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.659, ANCOVA; LSM difference = -0.16, 95% CI 2-sided [-0.87 to 0.55]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen 250 mg+Acetaminophen 500 mg; WSTD 0-6 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p < 0.001, ANCOVA; LSM difference = 2.62, 95% CI 2-sided [1.16 to 4.08]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Ibuprofen 250 mg; WSTD 0-6 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.135, ANCOVA; LSM difference = 0.79, 95% CI 2-sided [-0.25 to 1.82]
Statistical Analysis 15: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Acetaminophen 500 mg; WSTD 0-6 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.186, ANCOVA; LSM difference = 0.70, 95% CI 2-sided [-0.34 to 1.74]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg; WSTD 0-6 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.014, ANCOVA; LSM difference = 1.83, 95% CI 2-sided [0.37 to 3.29]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen 500 mg; WSTD 0-6 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.011, ANCOVA; LSM difference = 1.92, 95% CI 2-sided [0.45 to 3.39]
Statistical Analysis 18: Comparison: Ibuprofen 250 mg vs Acetaminophen 500 mg; WSTD 0-6 hours; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.865, ANCOVA; LSM difference = -0.09, 95% CI 2-sided [-1.12 to 0.94]

3. Secondary Outcome: Time to Return to Normal Body Temperature
Description: Time to return to normal body temperature was defined as time from initial measurement of normal body temperature (at baseline; before administration of first test dose of RSE to induce pyrexia) till the time at which normal temperature was achieved again after pyrexia. Normal body temperature was defined as the last non-missing body temperature value, assessed prior to or at the time of first RSE test dose.
Time Frame: Baseline (pre-dose) up to 8 hours post dose
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen 250 mg+Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 500 mg
Number analyzed (Participants) | 27 | 81 | 83 | 82
minutes | 360 [300 to 390] | 330 [240 to 360] | 390 [300 to 420] | 330 [270 to 360]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg+Acetaminophen 500 mg; Test type: Superiority; p = 0.449, Log Rank — Generalized log-rank test based on interval-censored survival analysis using nonparametric survival method
Statistical Analysis 2: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Ibuprofen 250 mg; Test type: Superiority; p = 0.142, Log Rank — Generalized log-rank test based on interval-censored survival analysis using nonparametric survival method
Statistical Analysis 3: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Acetaminophen 500 mg; Test type: Superiority; p = 0.822, Log Rank — Generalized log-rank test based on interval-censored survival analysis using nonparametric survival method
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; Test type: Superiority; p = 0.671, Log Rank — Generalized log-rank test based on interval-censored survival analysis using nonparametric survival method
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 500 mg; Test type: Superiority; p = 0.514, Log Rank — Generalized log-rank test based on interval-censored survival analysis using nonparametric survival method
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 500 mg; Test type: Superiority; p = 0.191, Log Rank — Generalized log-rank test based on interval-censored survival analysis using nonparametric survival method

4. Secondary Outcome: Time to Rescue Medication
Description: Time to rescue medication (other than study treatment) (in minutes) was defined as time from first dosing of study medication to the time a participant first takes a rescue medication, or to the end of the study time for participants that do not take any rescue medication prior to the end of the study. The rescue medication was defined as medication received for the treatment of fever during the time period from the administration of study medication to the time of end of the study.
Time Frame: 0 to 8 hours post dose
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen 250 mg+Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 500 mg
Number analyzed (Participants) | 27 | 81 | 83 | 82
minutes | NA [NA to NA] — Median, lower and upper limit of 95% CI was not estimable due to the low number of participants who had rescue medication. | NA [NA to NA] — Median, lower and upper limit of 95% CI was not estimable due to the low number of participants who had rescue medication. | NA [NA to NA] — Median, lower and upper limit of 95% CI was not estimable due to the low number of participants who had rescue medication. | NA [NA to NA] — Median, lower and upper limit of 95% CI was not estimable due to the low number of participants who had rescue medication.
Statistical Analysis 1: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Ibuprofen 250 mg; Test type: Superiority; p = 0.997, hazard ratio — P-value, hazard ratio (HR) and corresponding 95% CI were calculated based on the proportional hazards (PH) model with treatment term in the model
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg; Test type: Superiority; p = 0.998, Hazard Ratio — P-value, HR and corresponding 95% CI were calculated based on the PH model with treatment term in the model
Statistical Analysis 3: Comparison: Ibuprofen 250 mg vs Acetaminophen 500 mg; Test type: Superiority; p = 0.997, Hazard Ratio — P-value, HR and corresponding 95% CI were calculated based on the PH model with treatment term in the model

5. Secondary Outcome: Time Weighted Sum of Temperature Difference From 6 to 8 Hours
Description: WSTD 6-8 was defined as time-weighted sum of temperature differences between 6 to 8 hours post-dose, weighted by time elapsed between each 2 consecutive time points within 6 to 8 hours (6.5, 7, 7.5 and 8 hours). Temperature difference was defined as temperature at 6 hours minus the temperature at specified time points (6.5, 7, 7.5 and 8 hours).
Time Frame: 6 to 8 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees fahrenheit
Arm/Group | Placebo | Ibuprofen 250 mg+Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 500 mg
Number analyzed (Participants) | 27 | 81 | 83 | 82
degrees fahrenheit | 4.96 (2.228) | 5.69 (1.904) | 5.49 (2.261) | 5.84 (2.328)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg+Acetaminophen 500 mg; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.101, ANCOVA; LSM difference = 0.67, 95% CI 2-sided [-0.13 to 1.48]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Ibuprofen 250 mg; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.582, ANCOVA; LSM difference = 0.16, 95% CI 2-sided [-0.41 to 0.73]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg+Acetaminophen 500 mg vs Acetaminophen 500 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.614, ANCOVA; LSM difference = 0.15, 95% CI 2-sided [-0.43 to 0.72]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.212, ANCOVA; LSM difference = 0.51, 95% CI 2-sided [-0.29 to 1.32]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 500 mg; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.202, ANCOVA; LSM difference = 0.53, 95% CI 2-sided [-0.28 to 1.34]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 500 mg; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.965, ANCOVA; LSM difference = -0.01, 95% CI 2-sided [-0.58 to 0.55]

6. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between first dose of study drug and up to 24 hours after discharge (up to 32 hours) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 24 hours after discharge (up to 32 hours)
Population: Safety analysis set included all participants who received study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ibuprofen 250 mg+Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 500 mg
Number analyzed (Participants) | 29 | 87 | 87 | 87
Participants | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 24 hours after discharge (up to 32 hours)
Description: Safety analysis set included all participants who received study medication.
Arm/Group | Placebo | Ibuprofen 250 mg+Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 500 mg
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/87 | 0/87 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/87 | 0/87 | 0/87
Other Adverse Events (participants affected / at risk) | 1/29 | 1/87 | 0/87 | 0/87
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Ibuprofen 250 mg+Acetaminophen 500 mg (N=87) | Ibuprofen 250 mg (N=87) | Acetaminophen 500 mg (N=87)
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT02761980/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT02761980/SAP_001.pdf